CLINICAL TRIAL: NCT04799717
Title: Game-based Telehealth Therapeutic Intervention in First Onset Psychosis
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Janai Venugopalakrishnan, Clinical Assistant Professor, Stanford University
Other Study IDs: 59698
Record Dates: First submitted 2021-02-12; First posted 2021-03-16 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Psychotic Disorders; Schizophrenia Spectrum Disorders
Keywords: Telehealth, Therapy, intervention; Video game, CBT-P
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Gaming session — Participants will be provided the option to play an online game with the clinician for the first half of the session through an online platform.

SUMMARY:
The goal is to provide combination of 2 hours of weekly game based telehealth therapeutic intervention along with CBT-P for children identified with first onset psychosis or to be clinically high risk for psychosis thus widening therapeutic services offered. Target outcome measures are improvement in clinical symptoms, treatment engagement, and reduced hospitalization rates.

DETAILED DESCRIPTION:
Patients with first onset psychosis or clinical high risk for psychosis often have significant functional decline affecting social, academic, and daily living skills. Given their constellation of new onset psychotic symptoms of paranoia, delusions, hallucinations, and additionally co-morbid anxiety, or depression, patients most often present with school refusal, social withdrawal, aggression, poor self-care, and treatment noncompliance. This leads to decline in quality of life for both patients and families, along with increased sick days, recurrent hospitalizations, residential treatment center admissions which aren't always covered by insurance. Families are often left with very little to intervene and they carry the long-term disease burden of a significant diagnosis in addition to pocketing out of network costs for therapy. Further clinical programs like intensive outpatient programs or partial hospitalization programs often reject candidates with psychosis due to severity of symptoms and low levels of engagement when compared to their counterparts. County services offering in home therapeutic support services like rehabilitation, family therapy, peer support and wrap around services do not apply to insured patients thus causing huge gap in need for services. Early treatment with therapy and medications in first onset psychosis is very valuable as repeatedly shown clinically and in research.

Method: 10 patients in the 10-18 year age group meeting criteria for clinical high risk psychosis and schizophrenia spectrum disorders will be selected using DSM 5 criteria. Patients will be seen twice weekly for 15 weeks. They will be offered weekly individual telehealth therapy using game-based approach for first half of their visit to encourage engagement with therapist. Safe online videogames of their choice will be chosen, allowing usage of computer or electronics during session as needed to serve treatment purposes. The other half of the visit will focus on psychoeducation and utilizing CBT-P components targeting symptoms of psychosis. Patients will be assessed once a month clinically by treating psychiatrist in INSPIRE clinic to track symptom reduction, treatment engagement and hospitalization. Outcome measures will be tracked each month and data compiled between 4/2021-6/2021.

ELIGIBILITY:
Inclusion criteria is one of the following diagnoses:

* Clinical Diagnosis of Schizophrenia spectrum disorders
* Major Depressive Disorder with Psychotic Features
* Schizophrenia,
* Attenuated psychosis syndrome,
* Brief psychotic disorder,
* Schizoaffective Disorder,
* Schizophreniform disorder
* Unspecified psychotic disorder
* Clinical high risk for psychosis

Exclusion Criteria:

-Clinical Diagnosis of Intellectual Disability

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents and young adults ages 10 to 18 years of age with a psychotic disorder diagnosis or report of transient positive symptoms of psychosis that has lasted more than one week over the past year.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Hospitalization | The 15 week participation period
  Review patient's medical record for number of hospitalizations due to psychotic disorder
Patient Session Engagement | The 15 week participation period.
  Measure client engagement in treatment by providing a post-session survey. The survey has four questions to solicit client feedback on the therapy session. The clients will answer on a scale of 1-10 with 1 being the lowest and 10 being the highest score. Add all four numbers together to obtain the total score.
Brief Psychiatric Rating Scale Scores | The 15 week participation period.
  Perform the Brief Psychiatric Rating Scale (BPRS). The BPRS is a 21 questionaire of present of mental health symptoms wtih each question scored on a Likert scale of 1-7. A score of 01reflects that a particular question was not assessed and a score of 7 is highest severity of the symptom listed in each individual question. A total score is not calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Janani Venugopalakrishnan, MD MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford Universtiy, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrari M, McIlwaine SV, Reynolds JA, Archie S, Boydell K, Lal S, Shah JL, Henderson J, Alvarez-Jimenez M, Andersson N, Boruff J, Nielsen RKL, Iyer SN. Digital Game Interventions for Youth Mental Health Services (Gaming My Way to Recovery): Protocol for a Scoping Review. JMIR Res Protoc. 2020 Jun 24;9(6):e13834. doi: 10.2196/13834. PMID 32579117
- [Background] Landa Y, Mueser KT, Wyka KE, Shreck E, Jespersen R, Jacobs MA, Griffin KW, van der Gaag M, Reyna VF, Beck AT, Silbersweig DA, Walkup JT. Development of a group and family-based cognitive behavioural therapy program for youth at risk for psychosis. Early Interv Psychiatry. 2016 Dec;10(6):511-521. doi: 10.1111/eip.12204. Epub 2015 Jan 13. PMID 25585830
- [Background] Peters E, Crombie T, Agbedjro D, Johns LC, Stahl D, Greenwood K, Keen N, Onwumere J, Hunter E, Smith L, Kuipers E. The long-term effectiveness of cognitive behavior therapy for psychosis within a routine psychological therapies service. Front Psychol. 2015 Oct 29;6:1658. doi: 10.3389/fpsyg.2015.01658. eCollection 2015. PMID 26579041
- [Background] Rasskazova, Elena & Friedberg, Robert. (2016). CBT for psychosis prevention and treatment in youth. Current Psychiatry Reviews. 12.
- [Background] Stafford MR, Jackson H, Mayo-Wilson E, Morrison AP, Kendall T. Early interventions to prevent psychosis: systematic review and meta-analysis. BMJ. 2013 Jan 18;346:f185. doi: 10.1136/bmj.f185. PMID 23335473
- [Background] Stafford MR, Mayo-Wilson E, Loucas CE, James A, Hollis C, Birchwood M, Kendall T. Efficacy and safety of pharmacological and psychological interventions for the treatment of psychosis and schizophrenia in children, adolescents and young adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 11;10(2):e0117166. doi: 10.1371/journal.pone.0117166. eCollection 2015. PMID 25671707
- [Background] Stain HJ, Bucci S, Baker AL, Carr V, Emsley R, Halpin S, Lewin T, Schall U, Clarke V, Crittenden K, Startup M. A randomised controlled trial of cognitive behaviour therapy versus non-directive reflective listening for young people at ultra high risk of developing psychosis: The detection and evaluation of psychological therapy (DEPTh) trial. Schizophr Res. 2016 Oct;176(2-3):212-219. doi: 10.1016/j.schres.2016.08.008. Epub 2016 Aug 20. PMID 27554197
- [Background] Adery LH, Ichinose M, Torregrossa LJ, Wade J, Nichols H, Bekele E, Bian D, Gizdic A, Granholm E, Sarkar N, Park S. The acceptability and feasibility of a novel virtual reality based social skills training game for schizophrenia: Preliminary findings. Psychiatry Res. 2018 Dec;270:496-502. doi: 10.1016/j.psychres.2018.10.014. Epub 2018 Oct 9. PMID 30326433
- [Background] Yang CY, Lee TH, Lo SC, Beckstead JW. The effects of auditory hallucination symptom management programme for people with schizophrenia: a quasi-experimental design. J Adv Nurs. 2015 Dec;71(12):2886-97. doi: 10.1111/jan.12754. Epub 2015 Aug 18. PMID 26283291
- [Background] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167